CLINICAL TRIAL: NCT00533741
Title: Phase I, Double-Blinded, Placebo-Controlled Dosage Escalation Study of the Safety and Immunogenicity of Adjuvanted and Non-Adjuvanted Inactivated SARS Coronavirus (SARS-CoV) Vaccine Administered by the Intramuscular Route
Brief Title: SARS Coronavirus Vaccine (SARS-CoV)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-0021
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2010-03

CONDITIONS: Coronavirus (SARS-CoV)
Keywords: Severe Acute Respiratory Syndrome, Coronavirus, vaccine
MeSH Terms: conditions — Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- 1c (10 mcg) (Experimental): 4 subjects randomized in a 1:3 fashion to receive a two dose regimen of placebo or vaccine with 10 mcg of antigen and no adjuvant.
  Interventions: Drug: Placebo; Biological: SARS-CoV
- 2 (dose comparison stage) (Experimental): 54 subjects (9 per vaccine group) randomized 1:1:1:1:1:1 to receive vaccines containing, 2.5, 5.0, or 10.0 mcg of antigen without adjuvant, or 2.5 or 5.0 mcg of antigen with Alum, or placebo.
  Interventions: Drug: Aluminum hydroxide; Drug: Placebo; Biological: SARS-CoV
- 1a (2.5 mcg) (Experimental): 7 subjects randomized in a 1:3:3 fashion to receive a 2 dose regimen of placebo, vaccine containing 2.5 mcg of antigen and no adjuvant, or 2.5 mcg of antigen and Alum adjuvant.
  Interventions: Drug: Aluminum hydroxide; Drug: Placebo; Biological: SARS-CoV
- 1b (5.0 mcg) (Experimental): 7 subjects randomized in a 1:3:3 fashion to receive a 2 dose regimen of placebo, vaccine containing 5.0 mcg of antigen and no adjuvant, or 5.0 mcg of antigen and Alum adjuvant.
  Interventions: Drug: Aluminum hydroxide; Drug: Placebo; Biological: SARS-CoV

INTERVENTIONS:
Drug: Aluminum hydroxide — Adjuvant; administered with SARS-CoV vaccine.
  Arms: 1a (2.5 mcg); 1b (5.0 mcg); 2 (dose comparison stage)
Drug: Placebo — Saline for injection.
Biological: SARS-CoV — Whole-virus vaccine, grown in certified Vero cells and doubly inactivated by treatment with formalin and ultraviolet light (UV). Supplied in liquid formulation in single dose vials with and without aluminum hydroxide as an adjuvant. Doses supplied without aluminum hydroxide will be 2.5, 5.0 and 10.0 mcg. Doses supplied with aluminum hydroxide adjuvant will be 2.5 and 5.0 mcg.

SUMMARY:
Severe acute respiratory syndrome (SARS) is a viral illness that affects the respiratory (breathing) system. The purpose of this study is to evaluate the safety and protective (immune) responses to different doses of a SARS vaccine given with or without an adjuvant. An adjuvant is a substance that may be added to a vaccine to improve the immune response so that less of the vaccine may need to be given. Study participants will include 72 volunteers, ages 18-40, living in the Houston, Texas area. The study will take place at Baylor College of Medicine. Participants will receive 2 injections of vaccine or placebo (substance made to look like the study vaccine but contains no medication) given 1 month apart. Participants will fill out a memory aid (diary) to document daily temperature and illness signs and symptoms for 7-9 days after each injection. During the 9 study visits, several blood samples will be collected. Participants will be in the study for up to 211 days, including screening.

DETAILED DESCRIPTION:
Severe acute respiratory disease (SARS) is a recently emerged infectious disease that was first recognized in Guangdong Province, China, in November of 2002. Efforts to prevent the spread of this virus stopped the epidemic in July, 2003, but over 8,000 cases had occurred and almost 800 people died. A new virus, a coronavirus, was shown to be the cause and it is believed to be a virus of bats that infected some animals that, in turn, infected people and they gave it to other people. While it is unlikely to again become epidemic, the virus is thought to be a risk for spread to humans if it was released intentionally by a terrorist group. For that reason, the U.S. government is developing vaccines and drugs for use if spread should occur again. This study will test the safety and protective responses to a vaccine against SARS made by a vaccine company for this study. This protocol concerns Phase I clinical testing of an inactivated, purified SARS Coronavirus (CoV) vaccine administered with and without aluminum hydroxide (Alum) adjuvant. The rationale for development of vaccines against SARS-CoV is to provide a means of control in the event a new SARS-CoV epidemic occurs or there is a deliberate release of the virus. Inactivated SARS-CoV vaccine has been shown to induce neutralizing antibodies that block binding of the virus to its receptor, ACE2. The primary objectives of the study are to assess: reactogenicity of escalating doses of adjuvanted and non-adjuvanted, inactivated SARS-CoV vaccine among healthy young adult subjects given their first intramuscular (IM) vaccinations with this vaccine; reactogenicity of a repeat IM administration of the same material to healthy young adult subjects one month later; and development and persistence of immune responses to escalating doses of adjuvanted and non-adjuvanted, inactivated SARS-CoV vaccine 1 and 5 months after the second ("booster") vaccination. The secondary objective of this study is to assess immune responses to each vaccine 1 month after a single dose. This is a single center, Phase I, out-patient study of the reactogenicity (tolerability and safety) and immunogenicity of escalating doses of an inactivated SARS-CoV vaccine with and without aluminum hydroxide as an adjuvant. Each vaccine will be injected as primary and booster vaccinations a month apart in the subject's non-dominant deltoid muscle. Participants will include 72 healthy males or non-pregnant, non-lactating females, 18-40 years old from the Houston, Texas area. The study will be conducted at Baylor College of Medicine in 2 sequential stages. This study consists of a preliminary dose-escalation stage (1.a, 1.b, and 1.c) followed by a dose comparison stage (2) as follows: Stage 1a (2.5 mcg), 7 subjects randomized in a 1:3:3 fashion to receive a 2 dose regimen of placebo, vaccine containing 2.5 mcg of antigen and no adjuvant, or 2.5 mcg of antigen and Alum adjuvant; Stage 1b (5.0 mcg), 7 subjects randomized in a 1:3:3 fashion to receive a 2 dose regimen of placebo, vaccine containing 5.0 mcg of antigen and no adjuvant, or 5.0 mcg of antigen and Alum adjuvant; Stage 1c (10.0 mcg), 4 subjects randomized in a 1:3 fashion to receive a 2 dose regimen of placebo or vaccine with 10 mcg of antigen and no adjuvant; Stage 2, 54 subjects (9 per vaccine group) randomized 1:1:1:1:1:1 to receive vaccines containing, 2.5, 5.0, or 10.0 mcg of antigen without adjuvant, or 2.5 or 5.0 mcg of antigen with Alum, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and communicate in written and spoken English.
* Judged to be able to provide informed consent and has signed informed consent form prior to study participation.
* Male or female between 18 and 40 years of age.
* Females of childbearing potential agree to practice adequate contraception for the entire study period.
* Good general health as confirmed by medical history, history-directed physical examination, and laboratory assessments within normal ranges established by Baylor College of Medicine.
* Availability for follow-up for six months after the first vaccination.
* Willing and able to comply with protocol requirements.

Exclusion Criteria:

* Clinically significant medical disorder found by medical history or physical exam.
* History of anaphylaxis or other significant adverse event following immunization.
* History of or planned exposure to small mammalian animals that are from Asia, or were previously housed with Asian counterparts.
* Pregnant or lactating female.
* Acute illness (cough, congestion, malaise, diarrhea, feverishness and/or oral temperature > 99.5 degrees Fahrenheit, etc.) within a week of planned vaccination.
* Use of an immunosuppressive or immunomodulatory drug such as greater than 5 mg/day of prednisone orally, or greater than 800 mcg/day of inhaled beclomethasone for 2 or more consecutive weeks within 3 months prior to the first vaccination.
* History of or current substance abuse, including alcohol (e.g., greater than or equal to 4 six-packs of beer or equivalent per week regularly).
* History of receiving blood or blood products in the previous three months, or anticipated over the six month study period.
* Vaccination with a live vaccine within 30 days of study vaccination, or a non-replicating, inactivated or subunit vaccine within 14 days of study vaccination, or planned during the study.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B surface antigen (HbsAg).
* Positive serology for severe acute respiratory disease (SARS) S protein if testing is done.
* Use of any investigational or unregistered drug or vaccine within 30 days before the first study vaccination, or planned use during the study.
* Autoimmune disease (e.g., lupus, rheumatoid arthritis), malignancy or tumor.
* Bleeding disorder by history, or thrombocytopenia.
* Diagnosis of schizophrenia, bipolar disease or other major psychiatric disorder.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, loxapine, thioridazine, molindone, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Plans to enroll in another study before study completion (six months).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Frequency and description of serious adverse events (SAEs). | 5 months after receipt of the booster dose of vaccine.
Frequency of significant increases in serum antibody to CoV S protein in Enzyme Linked Immunosorbent Assay (ELISA) and in neutralization tests, and increases in Geometric Mean Titers (GMT)s in sera. | Screening, 1 and 5 months after the booster dose of vaccine.
Frequency and severity of solicited injection site and systemic signs and symptoms and unsolicited adverse events (AE) / SAEs. | 1 month after receipt of the first and second doses of vaccine.

SECONDARY OUTCOMES:
Frequency of significant serum antibody increases and increases in Geometric Mean Titers (GMT)s, as measured in neutralizing antibody tests and an ELISA against SARS-CoV S protein. | Collected just before the first vaccination and at 1 month (just before booster).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas, United States